CLINICAL TRIAL: NCT01460563
Title: Effects of Valproic Acid and Magnesium Sulphate on Rocuronium Requirement and Postoperative Analgesia in Patients Undergoing Craniotomy for Cerebrovascular Surgery
Brief Title: Valproic Acid, Magnesium Sulphate, Rocuronium Requirement, Postoperative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kim Mihyun, clinical professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Mg_orfil
Record Dates: First submitted 2011-10-19; First posted 2011-10-27 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Cerebral Aneurysm
Keywords: craniotomy; sodium valproate; rocuronium
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mg_orfil (Experimental): patients preloaded with sodium valproate receives MgSO4 during the craniotomy.
  Interventions: Drug: Magnesium Sulfate
- control_orfil (Placebo Comparator): patients preloaded with sodium valproate receives 0.9% saline as placebo.
  Interventions: Drug: 0.9% saline
- control_no orfil (Placebo Comparator): patients not preloaded with sodium valproate receives 0.9% saline as placebo.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Magnesium Sulfate — MgSO4 infusion: 50mg/kg bolus followed by continuous infusion
  Other Names: MgSO4
  Arms: Mg_orfil
Drug: 0.9% saline — 0.9% saline as same dose as MgSO4 as placebo
  Other Names: NaCl
  Arms: control_orfil
Drug: 0.9% saline — 0.9% saline as same dose as MgSO4 as placebo
  Other Names: NaCl
  Arms: control_no orfil; control_orfil

SUMMARY:
The investigators hypothesized that valproic acid will increase rocuronium requirement and MgSO4 infusion would reduce requirement of muscle relaxant in craniotomy patients preloaded with sodium valproate.

DETAILED DESCRIPTION:
Magnesium sulfate (MgSO4) is known to reduce requirement of muscle relaxant.

ELIGIBILITY:
Inclusion Criteria:

* 18- 65 years
* American society of anesthesiology physical status 1,2
* scheduled for elective craniotomy for aneurysm clipping or for superficial temporal artery-middle cerebral artery anastomosis

Exclusion Criteria:

body mass index <18.5 or >24.9 kg m-2; neuromuscular, renal, cardiovascular or hepatic insufficiency; Glasgow coma scale (GCS) <15; allergy to the study drugs; medications influencing NDMRs; breast feeding; pregnancy; and preoperative epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Rocuronium | participants will be followed for the duration of the surgery, an expected average of 5.5 hours.
  Roc 0.15mg/kg is injected when train of four (TOF) becomes 2 which is measured with TOF-watch Sx. The total amount of Roc that injected is recorded.
  The intervals of each Roc 0.15mg/kg injection will also be recorded.

SECONDARY OUTCOMES:
hemodynamics | participants will be followed for the duration of the surgery, an expected average of 5.5 hours; postoperative 24 hour; postoperative 48 hour
  mean arterial pressure and heart rate is measured for the duration of the surgery, an expected average of 5.5 hours; postoperative 24 hour; postoperative 48 hour.
total amount of anesthetics | participants will be followed at the end of the surgery, an expected average of 5.5 hours after induction of anesthesia..
  total amount of propofol and remifentanil infused is measured.
Magnesium concentration | from the induction of anesthesia until end of the surgery
  serum Magnesium concentration is measured just prior to anesthetic drug administration, 3 hour after the induction of anesthesia, and at the end of the surgery.
side effects | participants will be followed for the duration of the surgery, an expected average of 5.5 hours; postoperative 24 hour; postoperative 48 hour.
  complicaton associated with MgSO4 including muscle weakness, hot flush, and nausea/ vomiting.
pain, nausea & vomiting, analgesics use, antiemetics use, nicardipine use | patients will be followed from the end of the operation until postoperativ 48 h
  Pain will be assessed using numeric rating scale at 6 h, 24 h, and 48 h postoperately.
  Cumulative dose of analgesics and nicardipine, incidence of nicardipine and antiemtics use during 48h postoperatively will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sanghwan Do, Doctor, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang hopital, Seongnam-si, Gyeonggi-do, South Korea